CLINICAL TRIAL: NCT04895787
Title: Augmented Benefits of Different Exercise Types to Enhance Skill Learning in People With Parkinson's Disease
Brief Title: Benefits of Different Exercise Types to Enhance Walking for PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202012147RIND
Record Dates: First submitted 2021-05-13; First posted 2021-05-20 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Parkinson Disease; Gait Disorders, Neurologic
Keywords: Parkinson's disease; Skill learning; Transcranial magnetic stimulation; Gait training; Aerobic exercise; Resistance exercise
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic | interventions — Gait; Exercise; RE1-silencing transcription factor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The researcher(s) who will conduct the outcome assessments will be masked from the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aerobic exercise group (AEX) (Experimental): Gait training followed by 20 minutes of moderate to high intensity aerobic exercise on a recumbent bicycle.
  Interventions: Behavioral: Gait + aerobic exercise
- Resistance exercise group (REX) (Experimental): Gait training followed by 20 minutes of resistance training targeting major muscle groups.
  Interventions: Behavioral: Gait + resistance exercises
- Conventional physical therapy group (CPT) (Active Comparator): Gait training followed by 20 minutes of conventional PT programs that do not involve aerobic or resistance exercise.
  Interventions: Behavioral: Gait + conventional physical therapy
- Control group (CON) (Active Comparator): Gait training followed by 20 minutes of rest (sitting on a chair and read magazines).
  Interventions: Behavioral: Gait + rest

INTERVENTIONS:
Behavioral: Gait + aerobic exercise — Following skill-based gait training, the participants in the AEX group will engage in 20 minutes of moderate to high intensity aerobic exercise on a recumbent bicycle. The participants will first perform a brief warm-up, followed by 20 minutes of moderate to high intensity aerobic exercise pedaling at 60-80 rpm with a target heart rate range between 60-70% of heart rate reserve (HRR). Given the potential of having autonomic dysfunction in this population, it has been suggested that a RPE scale between 14-17 is appropriate.
  Other Names: gait training and aerobic exercise on a recumbent bicycle
  Arms: Aerobic exercise group (AEX)
Behavioral: Gait + resistance exercises — Following skill-based gait training, the participants in the REX group will engage in resistance training, which will target major muscle groups important for daily activities. The resistance training will be provided with free weights or therabands at an intensity of 8-12 repetition maximum (RM). Each muscle group should be trained with 8-12 repetitions ranging from 1 to 3 sets with resting intervals provided between each set. The target RPE scale will be set between 14-17, and the training load will be progressively increased as the participants improved.
  Other Names: gait training and muscle strengthening exercise
  Arms: Resistance exercise group (REX)
Behavioral: Gait + conventional physical therapy — Following skill-based gait training, the participants in the CPT group will receive conventional physical therapy, which may include stretching exercise, balance training, or practice over-ground walking based on the participant's need.
  Other Names: gait training and conventional physical therapy
  Arms: Conventional physical therapy group (CPT)
Behavioral: Gait + rest — Following skill-based gait training, the participants will sit and rest on a chair.
  Other Names: gait training and rest
  Arms: Control group (CON)

SUMMARY:
Background: Gait disturbance is one of the most common complaints from patients with Parkinson's disease (PD). It is well-established that people with PD have motor learning impairments. To enhance motor learning, several methods have been recommended, such as sleep, non-invasive brain stimulation techniques, and aerobic exercise. To date, only 2 studies have investigated the effects of acute aerobic exercise on motor learning in people with PD. It is yet unclear whether adding aerobic exercise after multiple motor training sessions can enhance motor learning in people with PD. Additionally, most prior evidences utilized moderate to high intensity aerobic exercise to facilitate motor learning, it is yet unclear whether other types of exercise (e.g., resistance training) could induce similar beneficial effects. Therefore, this proposed project is specifically designed to investigate the effects of adding aerobic or resistance exercise after motor training. To take a step further, this project will also determine the patient characteristics who may benefit from the intervention.

Objectives: (1) To examine whether adding specific exercise after training can facilitate learning on patients with Parkinson's disease. (2) To determine the characteristics of participants who may benefit from these types of intervention approach.

Methods: A total of 76 participants with idiopathic PD diagnosed by neurologists will be recruited. All eligible participants will be randomized into one of the 4 groups: aerobic group (AEX), resistance group (REX), conventional PT group (CPT), and control group (CON). All participants will receive 12 sessions of gait training. All outcome measures will be assessed before the intervention (pre-test), after the 6th intervention session (mid-test), after all 12 intervention sessions (post-test), and 1-month after the intervention (follow-up test). All assessments will be performed by an independent research assistant who will be blinded to the group allocation of the participants. The primary outcome will be gait performance, and the secondary outcomes will include measurements of cognitive and behavioral functions. Additionally, transcranial magnetic stimulation will be used to examine the changes of corticomotor excitability associated with the interventions.

DETAILED DESCRIPTION:
Background: Gait disturbance is one of the most common complaints from patients with Parkinson's disease (PD). It is well-established that due to the dysfunction of the corticostriatal circuits, people with PD have motor learning impairments and may consequently influence the effects of rehabilitation. To enhance motor learning, several methods have been recommended, such as sleep, non-invasive brain stimulation techniques, and aerobic exercise. To date, only 2 studies have investigated the effects of acute aerobic exercise on motor learning in people with PD. These 2 studies were cross-sectional studies that only provided a single bout of aerobic exercise and followed the effects on motor learning for 7 days. It is yet unclear whether adding aerobic exercise after goal-based motor skill training for multiple training sessions, like a regular clinical treatment regimen, can boost up the speed of motor skill acquisition and enhance retention and transfer performances for people with PD. Additionally, most prior evidences utilized moderate to high intensity aerobic exercise to facilitate motor learning, it is yet unclear whether other types of exercise (e.g., resistance training) could induce similar beneficial effects. To the best of our knowledge, no study is specifically designed to compare the addictive effect of aerobic or resistance exercise on motor skill learning in people with PD. Therefore, this proposed project is specifically designed to answer the above questions. To take a step further, this project will also determine the patient characteristics who may benefit from the intervention.

Objectives: (1) To examine whether adding aerobic or resistance exercise after walking skill training can facilitate learning of the walking task on patients with Parkinson's disease. (2) To determine the characteristics of participants who may benefit from these types of intervention approach.

The first aim of this study is to investigate investigate the effects of adding aerobic or resistance exercise after gait training in people with PD. The second aim is to further determine the characteristics of participants who benefit from the proposed training program..

Methods: A total of 76 participants with idiopathic PD diagnosed by neurologists will be recruited. All eligible participants will be randomized into one of the 4 groups: aerobic group (AEX), resistance group (REX), conventional PT group (CPT), and control group (CON). All participants will receive one-on-one intervention sessions with a trained physical therapist. Each intervention sessions will last 60 minutes, which will include 30 minutes of treadmill training and an additional therapy based on group allocation. The participants will come to the lab for 12 training sessions spread across 4 to 6 weeks. All outcome measures will be assessed before the intervention (pre-test), after the 6th intervention session (mid-test), after all 12 intervention sessions (post-test), and 1-month after the intervention (follow-up test). All assessments will be performed by an independent research assistant who will be blinded to the group allocation of the participants. The primary outcome will be gait performance, and the secondary outcomes will include Montreal Cognitive Assessment test, Stroop Color-Word test, Unified Parkinson's Disease Rating Scale, Fatigue Severity Scale, Activities-Specific Balance Confidence Scale, Parkinson's Disease Questionnaire-39, New Freezing of Gait Questionnaire, Geriatric Depression Scale, finger sequence task, Timed Up and Go test, 5 times sit to stand test. Transcranial magnetic stimulation will be used to examine the changes of corticomotor excitability associated with the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's Disease
* Able to follow instructions to perform the tasks
* The Montreal Cognitive Assessment, MoCA ≥ 20
* Be able to walk independently with or without devices for at least 10 meters

Exclusion Criteria:

* Has deep brain stimulation or pacemaker implanted in their body
* A self-history of seizure
* A family-history of epilepsy
* Pregnancy
* Uncontrolled medical conditions
* Unstable cardiovascular diseases
* Has other neurological or psychological disorders in addition to Parkinson's Disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in gait performances | Four time points: pre-test (before intervention, 0 week), mid-test (after 6th intervention sessions, up to 2 weeks), post-test (after all intervention sessions, up to 4 weeks), follow-up test (one month after intervention, up to 8 weeks)
  The participants will be required to walk along a walkway with their comfortable walking speed, fastest walking speed and under dual task condition for 3 times each. The gait performances will be captured by the Physilog®5 system (Gait Up, Renens, Switzerland), which include two inertial sensors with built-in 3D accelerometers and gyroscopes.Gait performances in pretest, mid-test, post-test, and follow-up test will be evaluated, and the trend of changes will be determined.

SECONDARY OUTCOMES:
Change in Montreal Cognitive Assessment (MoCA) | Four time points: pre-test (before intervention, 0 week), mid-test (after 6th intervention sessions, up to 2 weeks), post-test (after all intervention sessions, up to 4 weeks), follow-up test (one month after intervention, up to 8 weeks)
  The MoCA will be used to evaluate general cognitive function of the participants. It evaluates several cognitive functions including attention, set-shifting, short-term memory, verbal fluency, calculation, orientation, digit span, conceptual thinking, and visuospatial processing skills. The total score of MoCA is 30 with a higher score indicating better cognitive function. The MoCA has good to excellent psychometric properties. MoCA will be assessed at pretest, mid-test, post-test, and follow-up test, and the trend of changes among these time points will be determined.
Change in the Stroop Color-Word test | Four time points: pre-test (before intervention, 0 week), mid-test (after 6th intervention sessions, up to 2 weeks), post-test (after all intervention sessions, up to 4 weeks), follow-up test (one month after intervention, up to 8 weeks)
  The Stroop Color-Word test will be used to evaluate the changes in executive functions in people with PD. The executive functions involved in the Stroop Color-Word test are selective attention, inhibition, and set-shifting. The Stroop Color-Word test comprises the congruent and incongruent testing conditions. The congruent condition is when the color ink of a word is coherent with the written color name, and the incongruent condition is when the color ink differs from the written color name (e.g., the word 'red' written in blue ink). The participants are instructed to read out the ink color of the word, but not the color word name, as accurately and as fast as possible within 45 seconds. The Stroop Color-Word test will be assessed at pretest, mid-test, post-test, and follow-up test, and the trend of changes among these time points will be determined.
Change in the Unified Parkinson's Disease Rating Scale (UPDRS) | Four time points: pre-test (before intervention, 0 week), mid-test (after 6th intervention sessions, up to 2 weeks), post-test (after all intervention sessions, up to 4 weeks), follow-up test (one month after intervention, up to 8 weeks)
  The Unified Parkinson's Disease Rating Scale (UPDRS) is a well-established and widely used rating tool for the evaluation of disease severity of PD. This study will only evaluate Part 3 of the scale - the motor disturbances of the patients. The total score ranges from 0 to 132 for Part 3 of the UPDRS with a lower score indicates less PD symptoms and a higher score suggests more severe in PD disease. Internal consistency and validity has been established to be excellent for UPDRS. UPDRS will be assessed at pretest, mid-test, post-test, and follow-up test, and the trend of changes among these time points will be determined.
Change in fatigue severity questionnaire (FSS) | Four time points: pre-test (before intervention, 0 week), mid-test (after 6th intervention sessions, up to 2 weeks), post-test (after all intervention sessions, up to 4 weeks), follow-up test (one month after intervention, up to 8 weeks)
  The FSS will be used to determine how fatigue interferes an individual's daily living and social participation. It contains 9 items, and each item is scored on a 7-point scale with a score 1 indicates strongly disagree and score 7 indicates strongly agree. The total score ranges from 9 to 63, with a higher score indicate greater fatigue severity. FSS will be assessed at pretest, mid-test, post-test, and follow-up test, and the trend of changes among these time points will be determined.
Change in Activities-Specific Balance Confidence (ABC) Scale | Four time points: pre-test (before intervention, 0 week), mid-test (after 6th intervention sessions, up to 2 weeks), post-test (after all intervention sessions, up to 4 weeks), follow-up test (one month after intervention, up to 8 weeks)
  The Activities-Specific Balance Confidence (ABC) scale will be used to examine an individual's confidence level of not falling when performing activities of daily living. The ABC Scale contains 16 different activities performed indoors and outdoors. The participants will be asked to rate their confidence level (range from 0% to 100% of confidence) of not falling for each item. An average score of the 16 items (range from 0% to 100%) will be calculated to determine the participant's confidence level of not falling when performing the activities of daily living. The internal consistency and test-retest reliability of the ABC scale in patients with PD were excellent. The ABC scale will be assessed at pretest, mid-test, post-test, and follow-up test, and the trend of changes among these time points will be determined.
Change in Parkinson's Disease Questionnaire-39 (PDQ-39) | Four time points: pre-test (before intervention, 0 week), mid-test (after 6th intervention sessions, up to 2 weeks), post-test (after all intervention sessions, up to 4 weeks), follow-up test (one month after intervention, up to 8 weeks)
  The PDQ-39 is a self-report questionnaire containing 39 items assessing the impact of PD on quality of life. The PDQ-39 covers 8 dimensions: mobility, activities of daily living, emotional well-being, stigma, cognition, communication, and bodily discomfort. The participants are required to answer the questions based on their experiences in the preceding month prior to the interview. The scoring system for each item ranges from 0 (never have difficulty) to 4 (always have difficulty) with lower scores suggesting better quality of life. PDQ-39 will be assessed at pretest, mid-test, post-test, and follow-up test, and the trend of changes among these time points will be determined.
Change in New Freezing of Gait Questionnaire (NFOG-Q) | Four time points: pre-test (before intervention, 0 week), mid-test (after 6th intervention sessions, up to 2 weeks), post-test (after all intervention sessions, up to 4 weeks), follow-up test (one month after intervention, up to 8 weeks)
  The NFOG-Q will be used to evaluate the freezing frequency and severity of the patients with PD. It composes of 3 parts; in the first part, a video clip will be shown to the participants with PD and help to classify whether an individual is a freezer or non-freezer. The second and third part of the questionnaire is designed for freezers only. PartⅡassesses the severity of FoG according to the frequency and duration of the freezing episodes, while PartⅢevaluates the impact of freezing on daily activities, such as walking. The reliability and internal consistency of the NFOG-Q have been well-established for patients with PD. NFOG-Q will be assessed at pretest, mid-test, post-test, and follow-up test, and the trend of changes among these time points will be determined.
Change in Geriatric Depression Scale (GDS) | Four time points: pre-test (before intervention, 0 week), mid-test (after 6th intervention sessions, up to 2 weeks), post-test (after all intervention sessions, up to 4 weeks), follow-up test (one month after intervention, up to 8 weeks)
  The GDS is a self-report measure of depression in older adults. The GDS contains 15 items, and the users respond in a "Yes/No" format to each question in reference to the past 1 week. GDS will be assessed at pretest, mid-test, post-test, and follow-up test, and the trend of changes among these time points will be determined.
Change in The Timed Up and Go (TUG) Test | Four time points: pre-test (before intervention, 0 week), mid-test (after 6th intervention sessions, up to 2 weeks), post-test (after all intervention sessions, up to 4 weeks), follow-up test (one month after intervention, up to 8 weeks)
  The participants will initially sit on a comfortable chair with hips and knees flexed at 90°. Upon a 'GO' signal, the participants will stand up from the chair, walk for 3 meters, turn around, walk back to the chair, and sit down. The participants will be instructed to complete the task at their preferred/ comfortable speed. Good to excellent test-retest reliability and inter-rater reliability have been established in people with PD. TUG will be assessed at pretest, mid-test, post-test, and follow-up test, and the trend of changes among these time points will be determined.
Change in Five Times Sit-to-Stand (FTSTS) Test | Four time points: pre-test (before intervention, 0 week), mid-test (after 6th intervention sessions, up to 2 weeks), post-test (after all intervention sessions, up to 4 weeks), follow-up test (one month after intervention, up to 8 weeks)
  The FTSTS test will be evaluated to represent the strength and endurance of the lower limbs. The participants will be sat on a standardized chair, and they will be required to stand up and then sit down for 5 times as fast as possible. The amount of time the participants need to complete the task will be recorded, and a lesser amount of times would indicate better strength of the lower extremities. FTSTS will be assessed at pretest, mid-test, post-test, and follow-up test, and the trend of changes among these time points will be determined.
Change in motor evoked potential (MEP) | Four time points: pre-test (before intervention, 0 week), mid-test (after 6th intervention sessions, up to 2 weeks), post-test (after all intervention sessions, up to 4 weeks), follow-up test (one month after intervention, up to 8 weeks)
  Transcranial magnetic stimulation (TMS) will be used to evaluate the MEP. Peak-to-peak MEP amplitude is an indicator of the integrity and excitability of the corticospinal tract. MEP will be assessed at pretest, mid-test, post-test, and follow-up test, and the trend of changes among these time points will be determined.
Change in cortical silent period (CSP) | Four time points: pre-test (before intervention, 0 week), mid-test (after 6th intervention sessions, up to 2 weeks), post-test (after all intervention sessions, up to 4 weeks), follow-up test (one month after intervention, up to 8 weeks)
  Transcranial magnetic stimulation (TMS) will be used to evaluate the CSP. The CSP is a period when EMG activity being suppressed for a few hundred milliseconds after the MEP, and has often been used as an indicator of the inhibitory mechanism occurs within the corticospinal tract. CSP will be assessed at pretest, mid-test, post-test, and follow-up test, and the trend of changes among these time points will be determined.
Change in intracortical inhibition and facilitation | Four time points: pre-test (before intervention, 0 week), mid-test (after 6th intervention sessions, up to 2 weeks), post-test (after all intervention sessions, up to 4 weeks), follow-up test (one month after intervention, up to 8 weeks)
  Paired pulse TMS will be used to evaluate the intracortical inhibition and facilitation. Intracortical inhibition and facilitation will be assessed at pretest, mid-test, post-test, and follow-up test, and the trend of changes among these time points will be determined.
Change in muscle strength of lower extremity muscles | Four time points: pre-test (before intervention, 0 week), mid-test (after 6th intervention sessions, up to 2 weeks), post-test (after all intervention sessions, up to 4 weeks), follow-up test (one month after intervention, up to 8 weeks)
  Hand-held dynamometer will be used to measure changes in muscle strength. The muscle groups in interest are hip flexors and extensors, knee flexors and extensors, and ankle dorsiflexors. Measurement of each muscle group will be repeated 3 times and an average score will be recorded. Muscle strength will be assessed at pretest, mid-test, post-test, and follow-up test, and the trend of changes among these time points will be determined.
Change in six-minute walk test (6MWT) | Four time points: pre-test (before intervention, 0 week), mid-test (after 6th intervention sessions, up to 2 weeks), post-test (after all intervention sessions, up to 4 weeks), follow-up test (one month after intervention, up to 8 weeks)
  The 6MWT will be used to measure the muscle endurance and cardiopulmonary function of the participants. The participants will be required to walk back and forth along a 30-meter walkway continuously for 6 minutes. Participants will be instructed to walk as far as possible within the 6 minutes. If they are too tired to continue walking, they will be allowed to rest as needed but resume walking as soon as possible. Total distance that the participants walk will be recorded. Additionally, heart rate and RPE will also be recorded immediately after the test. The 6MWT will be assessed at pretest, mid-test, post-test, and follow-up test, and the trend of changes among these time points will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Yun Lee, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University, Taipei, Taiwan